CLINICAL TRIAL: NCT06365905
Title: Non-Invasive Identification of Endometrial Cancer/Endometrial Atypical Hyperplasia With an AI-Based Classifier Applied to Transvaginal Ultrasound in Patients With Post-Menopausal Bleeding
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-011680; NCI-2024-02550 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-011680 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo a transvaginal ultrasound examination and endometrial sampling per standard of care and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study evaluates if AI can be used with transvaginal ultrasound images for early detection of endometrial cancer or premalignant lesions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Prospective validation of an artificial intelligence (AI) algorithm applied to transvaginal ultrasound (TVUS) to identify patients with premalignant/malignant in a population of women with postmenopausal bleeding (PMB).

OUTLINE: This is an observational study.

Patients undergo a transvaginal ultrasound examination and endometrial sampling per standard of care and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years
* At least one episode of postmenopausal bleeding (PMB)
* Endometrial biopsy available from at Mayo Clinic (MN, AZ, FL), Mayo Clinic Health System (MCHS), or an external institution
* Acceptance to participate in the study

Exclusion Criteria:

* Diagnostic tests performed more than 90 days apart
* Physical impediment/refusal to undergo transvaginal ultrasound (TVUS)

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with at least one episode of postmenopausal bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of artificial intelligence (AI) algorithm applied to transvaginal ultrasound (TVUS) | Baseline
  Two static TVUS images (one longitudinal, one transversal) will be independently validated and compared to results of endometrial sampling. Outcomes from these will be compared with predictions made by the AI models for accuracy of assessing premalignant/malignant disease.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen E Glaser, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials